CLINICAL TRIAL: NCT02737917
Title: EmergeNcy Department Apneic Oxygenation Versus Usual Care During Rapid Sequence Intubation : A Randomized Controlled Trial (The ENDAO Trial)
Brief Title: EmergeNcy Department Apneic Oxygenation Versus Usual Care During Rapid Sequence Intubation
Acronym: ENDAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #16-003
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Diffuse Apneic Oxygenation
MeSH Terms: interventions — Oxygen; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diffuse apneic oxygenation (Experimental): This group of patients will receive the standard of care treatment of rapid sequence intubation (pre-oxygenation, induction and intubation) plus the application of oxygen.
  Interventions: Other: Oxygen; Other: Standard of care
- Usual care (Other): This group of patients will receive the standard of care treatment of rapid sequence intubation (pre-oxygenation, induction and intubation)
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Oxygen — 15 L of oxygen will be delivered to the patient by nasal cannula during the apnea period of rapid sequence intubation.
  Arms: Diffuse apneic oxygenation
Other: Standard of care — Rapid sequence intubation

SUMMARY:
To determine the impact, if any the application of oxygen during the apnea period of rapid sequence intubation has on patients being intubated in the emergency department.

DETAILED DESCRIPTION:
Hypoxia may occur during rapid sequence intubation (RSI) of emergency department patients (1-4). This condition may increase the risk of the patient suffering a cardiac arrest secondary to securing the airway. A part of RSI is pre-oxygenation, which is defined as placing the patient on 100% fraction of inspired O2 for 3 minutes prior to administering the induction agents (i.e. sedative and neuromuscular blocker) in order to increase the amount of oxygen present in the functional residual capacity of the patients lungs to prolong oxygen saturating during the apneic period of endotracheal intubation (5-9). In the last decade, physicians have developed a process known as diffuse apneic oxygenation (DAO) in order to mitigate the risk of oxygen desaturation during this apneic period. The process entails leaving the patient on high flow nasal cannula (HFNC) oxygen during the act of visualizing the vocal cords and placing the endotracheal tube. Over the years the practice has started to become more common in emergency departments, operating rooms and ICU's all over the world. Recently, a randomized controlled trial (called The FELLOW Trial) of this practice demonstrated no difference in desaturation rates between those patients that received DAO and those that did not (usual practice) in patients in the ICU (10). Some have commented that the findings of this study cannot be applied to emergency department patients, and so evidence is lacking in regards to this population.

Purpose of the study:

Although studies have started to investigate the efficacy of DAO in preventing desaturation during RSI, evidence is still lacking in the emergency department patient population. The primary question being asked is: does diffuse apneic oxygenation increase the average lowest arterial oxygen saturation during rapid sequence intubation when compared to usual care? Secondary question being asked is: does diffuse apneic oxygenation decrease the incidence of desaturation in general, as well as hypoxemia and severe hypoxemia? The third question being asked is: does diffuse apneic oxygenation increase the time to desaturation?

ELIGIBILITY:
Inclusion Criteria:

Any patient greater than 18 years of age that presents to the Lincoln medical and Mental Health Center Emergency Department requiring endotracheal intubation.

Exclusion Criteria:

Patients will be excluded from the primary outcome analysis, but included in the intention to treat analysis for the secondary outcome if they are not pre-oxygenated to the standard RSI protocol of 3 minutes with 100% fraction of inspired oxygen (FiO2) by means of bag valve mask, HFNC and/or non-rebreather; patients will be excluded from the study in general if they are in cardiac or traumatic arrest or they are intubated without an apneic period (awake intubation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Scott, MD, Study Chair — NYCHHC/Lincoln
Locations (1):
- Lincoln Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available

REFERENCES:
- [Background] Jaber S, Amraoui J, Lefrant JY, Arich C, Cohendy R, Landreau L, Calvet Y, Capdevila X, Mahamat A, Eledjam JJ. Clinical practice and risk factors for immediate complications of endotracheal intubation in the intensive care unit: a prospective, multiple-center study. Crit Care Med. 2006 Sep;34(9):2355-61. doi: 10.1097/01.CCM.0000233879.58720.87. PMID 16850003
- [Background] Griesdale DE, Bosma TL, Kurth T, Isac G, Chittock DR. Complications of endotracheal intubation in the critically ill. Intensive Care Med. 2008 Oct;34(10):1835-42. doi: 10.1007/s00134-008-1205-6. Epub 2008 Jul 5. PMID 18604519
- [Background] Simpson GD, Ross MJ, McKeown DW, Ray DC. Tracheal intubation in the critically ill: a multi-centre national study of practice and complications. Br J Anaesth. 2012 May;108(5):792-9. doi: 10.1093/bja/aer504. Epub 2012 Feb 6. PMID 22315326
- [Background] De Jong A, Molinari N, Terzi N, Mongardon N, Arnal JM, Guitton C, Allaouchiche B, Paugam-Burtz C, Constantin JM, Lefrant JY, Leone M, Papazian L, Asehnoune K, Maziers N, Azoulay E, Pradel G, Jung B, Jaber S; AzuRea Network for the Frida-Rea Study Group. Early identification of patients at risk for difficult intubation in the intensive care unit: development and validation of the MACOCHA score in a multicenter cohort study. Am J Respir Crit Care Med. 2013 Apr 15;187(8):832-9. doi: 10.1164/rccm.201210-1851OC. PMID 23348979
- [Background] Baillard C, Fosse JP, Sebbane M, Chanques G, Vincent F, Courouble P, Cohen Y, Eledjam JJ, Adnet F, Jaber S. Noninvasive ventilation improves preoxygenation before intubation of hypoxic patients. Am J Respir Crit Care Med. 2006 Jul 15;174(2):171-7. doi: 10.1164/rccm.200509-1507OC. Epub 2006 Apr 20. PMID 16627862
- [Background] Mort TC. Preoxygenation in critically ill patients requiring emergency tracheal intubation. Crit Care Med. 2005 Nov;33(11):2672-5. doi: 10.1097/01.ccm.0000187131.67594.9e. PMID 16276196
- [Background] Mort TC, Waberski BH, Clive J. Extending the preoxygenation period from 4 to 8 mins in critically ill patients undergoing emergency intubation. Crit Care Med. 2009 Jan;37(1):68-71. doi: 10.1097/CCM.0b013e318192845e. PMID 19050620
- [Background] Vourc'h M, Asfar P, Volteau C, Bachoumas K, Clavieras N, Egreteau PY, Asehnoune K, Mercat A, Reignier J, Jaber S, Prat G, Roquilly A, Brule N, Villers D, Bretonniere C, Guitton C. High-flow nasal cannula oxygen during endotracheal intubation in hypoxemic patients: a randomized controlled clinical trial. Intensive Care Med. 2015 Sep;41(9):1538-48. doi: 10.1007/s00134-015-3796-z. Epub 2015 Apr 14. PMID 25869405
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Semler MW, Janz DR, Lentz RJ, Matthews DT, Norman BC, Assad TR, Keriwala RD, Ferrell BA, Noto MJ, McKown AC, Kocurek EG, Warren MA, Huerta LE, Rice TW; FELLOW Investigators; Pragmatic Critical Care Research Group. Randomized Trial of Apneic Oxygenation during Endotracheal Intubation of the Critically Ill. Am J Respir Crit Care Med. 2016 Feb 1;193(3):273-80. doi: 10.1164/rccm.201507-1294OC. PMID 26426458
- [Background] Ramachandran SK, Cosnowski A, Shanks A, Turner CR. Apneic oxygenation during prolonged laryngoscopy in obese patients: a randomized, controlled trial of nasal oxygen administration. J Clin Anesth. 2010 May;22(3):164-8. doi: 10.1016/j.jclinane.2009.05.006. PMID 20400000

RESULTS

PARTICIPANT FLOW:
Groups:
- Apneic Oxygenation: This group of patients will receive the standard of care treatment of rapid sequence intubation (pre-oxygenation, induction and intubation) plus the application of oxygen.
  Oxygen: 15 L of oxygen will be delivered to the patient by nasal cannula during the apnea period of rapid sequence intubation.
  Standard of care: Rapid sequence intubation
Period: Overall Study
Arm/Group | Apneic Oxygenation | Usual Care
Started | 103 | 103
Completed | 100 | 100
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apneic Oxygenation | Usual Care | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Full Range); unit: years] | 54.2 [21 to 89] | 55.1 [22 to 93] | 54.7 [21 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 58 | 59 | 117
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200
American Society of Anesthesia Classification [Mean (Full Range); unit: units on a scale] — The American Society of Anesthesia Classification is a scale system for assessing the fitness of patients before receiving anesthesia. Class 1 is a healthy person; Class 2 is mild systemic disease; Class 3 is severe systemic disease; Class 4 is Severe systemic disease that is a constant threat to life. 1 is the best and 4 is the worst.
  units on a scale | 2.67 [1 to 4] | 2.69 [1 to 4] | 2.68 [1 to 4]
Cormack-Lehane Grade/Scale of View [Mean (Full Range); unit: units on a scale] — The Cormack-Lehane Grade View is a scale from 1 to 4 (1,2,3,4) that numerical represent the view of the vocal cords during intubation. A lower number equates to the better view (i.e. 1=full view of the vocal cords) and higher numbers a worse view (i.e. 4=no view of the vocal cords).
  units on a scale | 1.41 [1 to 4] | 1.48 [1 to 4] | 1.44 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Mean (Average) Arterial Oxygen Saturation
Description: the average oxygen saturation as measured by peripheral capillary oxygen saturation (SpO2)
Time Frame: within 2 minutes of confirmation of endotracheal tube placement
Measure: Mean (95% Confidence Interval); unit: Percent Saturation (SpO2)
Arm/Group | Apneic Oxygenation | Usual Care
Number analyzed (Participants) | 100 | 100
Percent Saturation (SpO2) | 92 [91 to 93] | 93 [92 to 94]

2. Secondary Outcome: Rates of Desaturation
Description: number of patients per group that desaturated to less than 90% and less than 80%
Time Frame: within 2 minutes of confirmation of endotracheal tube placement
Population: All patients undergoing rapid sequence intubation receiving either Apneic Oxygenation or Usual Care
Measure: Count of Participants; unit: Participants
Arm/Group | Apneic Oxygenation | Usual Care
Number analyzed (Participants) | 100 | 100
Participants
  Desaturation >=80% | 17 | 15
  Desaturation <80% | 3 | 4
  No Desaturation to <90% or 80% | 80 | 81

ADVERSE EVENTS:
Time Frame: 30 days
Description: Serious adverse events (peri-intubation cardiac arrest, bradycardia) are related to hypoxemia during endotracheal intubation in general but not known to occur due to the administration of supplemental oxygen during such procedure.
Arm/Group | Apneic Oxygenation | Usual Care
All-Cause Mortality (participants affected / at risk) | 14/100 | 16/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes